CLINICAL TRIAL: NCT07231393
Title: Evaluation of Observation Periods and Biphasic Reaction Risk Factors in Pediatric Anaphylaxis Cases in the Pediatric Emergency Department: A Retrospective Study
Brief Title: Observation Periods and Biphasic Reaction Risk Factors in Pediatric Emergency Anaphylaxis Cases
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Aykut Çağlar, MD, Assoc. Prof, Aydin Adnan Menderes University
Other Study IDs: ADUPEDANAPH
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Child; Anaphylaxis; Pediatric Emergency Care; Biphasic Anaphylactic Reaction
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Anaphylaxis Cohort: Children under 18 years of age who presented to the Pediatric Emergency Department of Adnan Menderes University Hospital between January 2014 and December 2024 with a diagnosis of anaphylaxis, defined according to WAO 2020 criteria. All patients meeting eligibility criteria were included retrospectively from medical records.

SUMMARY:
This study reviews the medical records of children who presented to the pediatric emergency department of Adnan Menderes University Hospital with a diagnosis of anaphylaxis between January 2014 and December 2024. The aim is to determine how long children were observed in the emergency department, how often biphasic reactions (a second wave of symptoms) occurred, and which risk factors (such as delayed adrenaline use or asthma) may increase this risk. The results will help improve the care of children with anaphylaxis and guide recommendations for safe observation times.

DETAILED DESCRIPTION:
Anaphylaxis is a severe, potentially life-threatening systemic hypersensitivity reaction with rapid onset. Its incidence in children has been rising worldwide. Although international recommendations emphasize the importance of post-reaction monitoring, the optimal observation period in pediatric patients remains uncertain, largely due to the risk of biphasic reactions, defined as recurrence of symptoms after initial resolution within 1-72 hours.

This retrospective observational study was conducted in the Pediatric Emergency Department of Adnan Menderes University Hospital. All patients younger than 18 years who presented with anaphylaxis between January 1, 2014, and December 31, 2024, were included. Diagnosis was based on the World Allergy Organization (WAO) 2020 criteria. Data were obtained from electronic medical records and emergency department charts.

Collected variables included demographics (age, sex), season of presentation, suspected triggers (food, drug, insect sting, exercise, idiopathic), clinical manifestations (cutaneous, respiratory, cardiovascular, gastrointestinal, neurological), comorbidities (such as asthma), acute treatments (epinephrine administration, time to first dose, number of doses, corticosteroids, antihistamines, fluid therapy), observation duration, need for hospital admission, and occurrence of biphasic reactions.

The primary objective is to determine the incidence and timing of biphasic reactions. Secondary objectives are to assess the average observation period in the emergency department, the frequency of hospital admission, and risk factors associated with biphasic reactions, including delayed epinephrine administration and history of asthma. Statistical analysis will include descriptive methods, group comparisons, and logistic regression to identify independent predictors of biphasic reactions.

This study is expected to contribute real-world data on pediatric anaphylaxis and inform clinical practice regarding safe observation times. Results will be compared with existing evidence and may support improvements in pediatric emergency protocols for anaphylaxis management.

ELIGIBILITY:
Inclusion Criteria:

Age <18 years

* Diagnosis of anaphylaxis according to World Allergy Organization (WAO) 2020 criteria
* Complete clinical data available in medical records

Exclusion Criteria:

* Incomplete or missing clinical data
* Cases not meeting WAO 2020 anaphylaxis definition
* Patients presenting with isolated urticaria or localized allergic reactions only

Ages: 0 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children and adolescents (<18 years) who presented to the Pediatric Emergency Department of Adnan Menderes University Hospital between January 1, 2014, and December 31, 2024, with a diagnosis of anaphylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2014-05; Primary Completion 2024-11 (Actual); Study Completion 2025-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Biphasic Reactions | Within 72 hours of the initial anaphylaxis episode
  he proportion of pediatric patients who developed a biphasic reaction, defined as recurrence of anaphylaxis symptoms after complete resolution of the initial episode, within 1-72 hours.

SECONDARY OUTCOMES:
Mean Observation Period in the Pediatric Emergency Department | During index visit (hours)
  Average length of observation (in hours) in the pediatric emergency department following initial anaphylaxis management.
Risk Factors Associated with Biphasic Reactions | During index visit and follow-up within 72 hours
  Identification of independent predictors for biphasic reactions (e.g., history of asthma, delayed epinephrine administration, initial clinical severity, need for multiple epinephrine doses).

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Çağlar, Principal Investigator — Aydın Adnan Menderes University Hospital, Department of Pediatric Emergency Care

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data. Summary results will be available in published articles.

REFERENCES:
- [Background] Soyak Aytekin E, Sirin S, Kiratli Nalbant E, Ata N, Sertcelik A, Ulgu MM, Birinci S, Harmanci K, Akelma Z. Changes in anaphylaxis trends and characteristics in emergency department admissions in Turkiye: From 2015 to 2021 based on the Ministry of Health database. World Allergy Organ J. 2024 Dec 24;18(1):101019. doi: 10.1016/j.waojou.2024.101019. eCollection 2025 Jan. PMID 39810830
- [Background] Gaspar A, Santos N, Faria E, Pereira AM, Gomes E, Camara R, Rodrigues-Alves R, Borrego LM, Carrapatoso I, Carneiro-Leao L, Morais-Almeida M, Delgado L, Pedro E, Branco-Ferreira M; Portuguese Society of Allergology and Clinical Immunology (SPAIC) Anaphylaxis Interest Group. Anaphylaxis in children and adolescents: The Portuguese Anaphylaxis Registry. Pediatr Allergy Immunol. 2021 Aug;32(6):1278-1286. doi: 10.1111/pai.13511. Epub 2021 Apr 18. PMID 33774834
- [Background] Muraro A, Worm M, Alviani C, Cardona V, DunnGalvin A, Garvey LH, Riggioni C, de Silva D, Angier E, Arasi S, Bellou A, Beyer K, Bijlhout D, Bilo MB, Bindslev-Jensen C, Brockow K, Fernandez-Rivas M, Halken S, Jensen B, Khaleva E, Michaelis LJ, Oude Elberink HNG, Regent L, Sanchez A, Vlieg-Boerstra BJ, Roberts G; European Academy of Allergy and Clinical Immunology, Food Allergy, Anaphylaxis Guidelines Group. EAACI guidelines: Anaphylaxis (2021 update). Allergy. 2022 Feb;77(2):357-377. doi: 10.1111/all.15032. Epub 2021 Sep 1. PMID 34343358
- [Background] Cardona V, Ansotegui IJ, Ebisawa M, El-Gamal Y, Fernandez Rivas M, Fineman S, Geller M, Gonzalez-Estrada A, Greenberger PA, Sanchez Borges M, Senna G, Sheikh A, Tanno LK, Thong BY, Turner PJ, Worm M. World allergy organization anaphylaxis guidance 2020. World Allergy Organ J. 2020 Oct 30;13(10):100472. doi: 10.1016/j.waojou.2020.100472. eCollection 2020 Oct. PMID 33204386

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-10-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT07231393/Prot_SAP_ICF_000.pdf